CLINICAL TRIAL: NCT03369782
Title: Effect of Neuromuscular Blockade on Surgical Conditions and Patient Reported Comfort Scores in Total Hip Replacement Arthroplasty
Brief Title: Effect of NMBA on Surgical Conditions in THR
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: refocusing of research priorities
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Dr. Alain Kalmar, MD, PhD, Staff Anesthetist, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMS.2017.033
Record Dates: First submitted 2017-12-04; First posted 2017-12-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Surgery; Postoperative Pain
Keywords: Muscle Tension; Skeletal Muscle Relaxants; Arthroplasties, Hip Replacement; Rocuronium; sugammadex
MeSH Terms: conditions — Pain, Postoperative | interventions — Rocuronium; Sugammadex; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Group A receives rocuronium, followed by sugammadex. Group B receives placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The syringes are prepared by the research assistant who was not involved in patient management. The anesthetist and surgeon are blinded for patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo alternative for rocuronium and for sugammadex
  Interventions: Drug: Placebo
- Rocuronium (Active Comparator): Rocuronium as bolus and in syringe pump Sugammadex just before reduction of the joint
  Interventions: Drug: Rocuronium; Drug: Sugammadex

INTERVENTIONS:
Drug: Rocuronium — rocuronium is administered in bolus and continuous infusion
  Other Names: Esmeron
  Arms: Rocuronium
Drug: Sugammadex — Sugammadex is administered just before reduction of the joint
  Other Names: Bridion
  Arms: Rocuronium
Drug: Placebo — Placebo is administered as alternative to rocuronium in a bolus and in a syringe pump.
  Placebo is administered as alternative to sugammadex
  Other Names: Saline 0.9%
  Arms: Placebo

SUMMARY:
During Total hip replacement arthroplasty (THA), the hip joint first must be luxated in order to have access to the joints. A lot of force and torque must be carried out on the joint to perform this manipulation. This is both difficult for the surgeon and may cause additional tissue damage and postoperative pain. After placement of the prosthesis and reduction of the joint, the tension of the hip joint must be evaluated by the surgeon to ascertain the adequacy of the prosthesis. During luxation, minimal muscle tension would be ideal, while after reduction of the joint, normal muscle tension is desired to permit assessment of the mechanics of the hip joint.

The aim of the study is to investigate whether deep neuromuscular block, combined with a reversal before mechanics assessment improves surgical conditions, surgical time, and postoperative patient comfort.

DETAILED DESCRIPTION:
2X20 patients are randomised: Rocuronium-group (R-group) and Placebo-group (P-group).

All patients receive standardised multimodal intravenous analgesia. After standardised induction of anasthesia and patient positioning, the patient is administered either placebo or rocuronium 0.9 mg/kg, followed by continuous infusion of either placebo or rocuronium 0.4 mg/kg/h. 1 minute before reduction of the hip joint, the patient is administered either sugammadex (R-group) or placebo (P-group) for full reversal of the neuromuscular block.

During the surgery, time points are recorded for: incision, start luxation of the joint, start reduction of the joint, start skin closure.

The surgeon is blinded for patient allocation. At three moments (after luxation, just before reduction of the joint, and after assessment of joint mechanics), the surgeon is asked to appraise the surgical conditions on an analogue scale.

Postoperative analgesic consumption and pain scores are recorded. VAS scores for knee pain and hip pain are assessed before surgery, at the moment of discharge from the post-anesthesia care unit (=D0), the morning after surgery (=D1), at D2, and at D7.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* eligible for primary THA
* BMI <35

Exclusion Criteria:

* neurological or psychiatric disorders
* intolerance or allergy against investigational drugs or any of the drugs used in the standardized analgetics scheme (acetaminophen, diclofenac, ketamine, clonidine, lidocaine)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-15 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Surgical conditions during luxation on a four-grade numeric scale | during surgery, during luxation of the joint
  Excellent - good but not optimal - poor but acceptable - unacceptable

SECONDARY OUTCOMES:
Patient reported pain scores on a VAS score (0-100 ; 0=no pain , 100=worst pain) | day 0-1-2-7 (day 0 = day of surgery)
  Patient reported pain scores in knee and hip after surgery at day 0-1-2-7
surgery time | during surgery
  time (in minutes) of surgery between incision and reduction, and between reduction and skin closure
Surgical conditions during reduction of the joint on a four-grade numeric scale | during surgery, during reduction of the joint
  Excellent - good but not optimal - poor but acceptable - unacceptable
Surgical conditions for assessment of joint kinetics on a four-grade numeric scale | during surgery, after reduction of the joint
  Excellent - good but not optimal - poor but acceptable - unacceptable

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, MD, PhD, MSc, Principal Investigator — Maria Middelares Hospital
Locations (1):
- AZ Maria Middelares, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
scores of surgical conditions patient-reported pain scores data about surgery time